CLINICAL TRIAL: NCT03588533
Title: Safety and Efficacy Evaluation of Capecitabine, Cisplatin, and Herzuma Combination Chemotherapy for the First Line Treatment of Advanced Gastric or Gastroesophageal Junction Adenocarcinoma Patients.
Brief Title: Herzuma-capecitabine/Cisplatin for Gastric Cancer
Acronym: HERZUMA-GC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sung Yong Oh (Other)
Collaborators: Celltrion (Industry)
Responsible Party: Sponsor-Investigator, Sung Yong Oh, Pricipal Investigator, Dong-A University Hospital
Organization: Dong-A University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAUHIRB-18-121
Record Dates: First submitted 2018-07-01; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: HER-2 Positive Gastric Cancer; Metastatic Cancer
Keywords: HER-2 Positive; Gastric or gastroesophageal adenocarcinoma; Herzuma
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Trastuzumab; Capecitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: * Herzuma 8mg/kg loading over 90min (1st cycle)
  * Herzuma 6mg/kg maintenance over 30min (2nd cycle~ ) every 3 weeks
  * Capecitabine 1000mg/m2 p.o. bid D1-D14 every 3 weeks
  * Cisplatin 60~100mg/m2 i.v. D1 every 3 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Herzuma-capecitabine/cisplatin(XP) (Experimental): * Trastuzumab (Herzuma) 8mg/kg loading over 90min (1st cycle)
  * Trastuzumab (Herzuma) 6mg/kg maintenance over 30min (2nd cycle~ ) every 3 weeks
  * Capecitabine 1000mg/m2 p.o. bid D1-D14 every 3 weeks
  * Cisplatin 60~100mg/m2 i.v. D1 every 3 weeks
  Interventions: Drug: Trastuzumab; Drug: Capecitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Trastuzumab — * Trastuzumab (Herzuma) 8mg/kg loading over 90min (1st cycle)
  * Trastuzumab (Herzuma) 6mg/kg maintenance over 30min (2nd cycle~ ) every 3 weeks
  Other Names: Herzuma
Drug: Capecitabine — - Capecitabine 1000mg/m2 p.o. bid D1-D14 every 3 weeks
  Other Names: Xeloda
Drug: Cisplatin — - Cisplatin 60~100mg/m2 i.v. D1 every 3 weeks

SUMMARY:
Stomach cancer is the fifth largest cancer in the world. Despite many combinations of studies, metastatic stomach cancer shows a median survival period of 10 to 12 months.

According to a report in Korea in 2010, 17 % of cancer patients had over-expression of human epidemiology growth factor receptor 2 (HER-2). And Using of Trastuzumab reported better results.Herzuma® is the Trastuzumab biosimilar (Biosimilar) cloned antibody.

In this study, the investigators want to prospectively analyze the effects and side effects of Herzuma® in gastric or gastroesophageal adenocarcinoma.

DETAILED DESCRIPTION:
Stomach cancer is the fifth largest cancer in the world, with an estimated 723,000 patients each year, and cancer-related deaths being the third leading cause. In contrast to the decline in the West, the Far East Asia, including South Korea, showed a high prevalence of cancer. In 2014, 29,854 new cases of cancer were reported in Korea. This is the second most important cancer in terms of incidence and the third in cancer related mortality.

The 5 year survival rate has increased to 74 % due to increased early detection of stomach cancer, but in the case of metastatic stomach cancer, the rate of gastric cancer is about one-third of the total number of stomach cancer cases, resulting in poor outcomes. Treatment is 5-fluorouracil, Oxaliplatin, Irinotecan, Epirubicin , Docetaxel, etc. based on platinum or non-platinum. Despite many combinations of studies, metastatic stomach cancer shows a median survival period of 10 to 12 months..

According to a report in Korea in 2010, 17 % of cancer patients had over-expression of human epidemiology growth factor receptor-2(HER-2). And Using of Trastuzumab reported better results in progression free survival (18.6 months vs. 17.1 months) and total overall survival (13.8 months vs. 11.1 months) (hazard ratio 0.74 ; 95 % confidential interval(CI) 0.60-0.91 ; p=0.0046) Trastuzumab was first used for HER-2 and breast cancer, and in three weeks of treatment, it is recommended to perform an induction phase of 8 mg/kg of 90 min and then a maintenance phase of 6mg/kg of 30min to 60min infusion. However, clinical research and data analysis are required because of concerns of toxic expression due to short-term injection. The phase I study of the maintenance 30 minutes toxicity was performed in breast cancer, and there was little difference from 60 minutes of injection in a 250ml or 100ml solution or new toxic event.

Herzuma® is the Trastuzumab biosimilar (Biosimilar) cloned antibody. In the phase I pharmacodynamics study, same the results with trastuzumab were reported. Biosimilar use was approved based on the results of a phase III clinical study on breast cancer. A double-blind, random assignment test was conducted on 549 HER-2 positive breast cancer patients comparing the validity and stability of Trastuzumab. The primary goal was to achieve a postoperative pathologic complete remission in 46.8 % of Herzuma® compared to 50.4% of trastuzumab. In addition, the secondary goal of "overall response rate " and "pharmacodynamics" showed the same results as the Trastuzumab control group.

Biosimilar Herzuma® licensed through breast cancer study also can be used in HER-2 overexpressed stomach cancer. However, there has not been a study on the effects and side effects of the drug.

So in this study, the investigators want to prospectively analyze the effects and side effects of Herzuma® in gastric or gastroesophageal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Gastric or gastroesophageal junction adenocarcinoma
2. HER-2 immuno-histochemical (IHC) (3 +) stain or her-2 silver in situ hybridization(SISH)/fluorescence in situ hybridization(FISH) (+)
3. Herzuma® -capecitabine/cisplatin combination regimen is planned as a first line treatment

Exclusion Criteria:

1. Other type of cancer of Gastric or gastroesophageal junction adenocarcinoma (e.g., lymphoma, sarcoma)
2. HER-2 (0/1+) in IHC or her-2 SISH/FISH (-).
3. Patients who previously performed stomach cancer treatment as a palliative setting.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-10 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Adverse event | up to 12 months
  Adverse event related with Herzuma

SECONDARY OUTCOMES:
Overall response rate | up to 6 months
  complete response+partial response by RECIST
Progression free survivals (PFS) | up to 12 months
  PFS
All adverse events | up to 12 months
  All adverse events during treatment
Overall survivals (OS) | up to 12 months
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Oh, MD, Principal Investigator — Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Busan, South Korea